CLINICAL TRIAL: NCT01496573
Title: Observational - CRKL Expression at the Protein Level in Rhabdomyosarcoma Tumors by Tissue Microarray (TMA)
Brief Title: Biomarkers in Tumor Tissue Samples From Younger Patients With Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST12B4; NCI-2012-00094 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-12-16; First posted 2011-12-21 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Alveolar Childhood Rhabdomyosarcoma; Childhood Rhabdomyosarcoma; Embryonal Childhood Rhabdomyosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Basic science (biomarker analysis): Archived tumor tissue samples are analyzed for CRKL expression.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies biomarkers in tumor tissue samples from younger patients with rhabdomyosarcoma. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate CRKL expression at the protein level in rhabdomyosarcoma tumors by tissue microarray (TMA).

OUTLINE:

Archived tumor tissue samples are analyzed for CRKL expression.

ELIGIBILITY:
Inclusion Criteria:

* Alveolar rhabdomyosarcoma and embryonal rhabdomyosarcoma specimens from the Children Oncology Group (COG) tumor microarrays (TMAs)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Alveolar rhabdomyosarcoma and embryonal rhabdomyosarcoma
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2011-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
CRKL expression at the protein level | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Lee Helman, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States